CLINICAL TRIAL: NCT00807807
Title: Phase III Study of the Effects of Folic Acid Supplementation on Serum Folate and Plasma Homocysteine in Older Adults: A Dose-Response Trial
Brief Title: Evaluating the Effects of Folic Acid Supplementation in Older Adults: The Folic Acid Supplementation Trial (The FAST Study)
Acronym: FAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Johns Hopkins University (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Lawrence J. Appel, MD, MPH, Johns Hopkins University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 617; U01HL050981 (NIH); M01RR000052 (NIH)
Record Dates: First submitted 2008-12-10; First posted 2008-12-12 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-12

CONDITIONS: Heart Diseases
Keywords: Plasma Homocysteine Concentration; Folate; Homocysteine; Supplements; Folic Acid
MeSH Terms: conditions — Heart Diseases | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator): Participants will receive placebo folic acid.
  Interventions: Drug: Placebo Folic Acid
- 2 (Experimental): Participants will receive 100 mcg of folic acid.
  Interventions: Dietary Supplement: Folic Acid
- 3 (Experimental): Participants will receive 400 mcg of folic acid.
  Interventions: Dietary Supplement: Folic Acid
- 4 (Experimental): Participants will receive 1000 mcg of folic acid.
  Interventions: Dietary Supplement: Folic Acid
- 5 (Experimental): Participants will receive 2000 mcg of folic acid.
  Interventions: Dietary Supplement: Folic Acid

INTERVENTIONS:
Dietary Supplement: Folic Acid — 100 mcg, 400 mcg, 1000 mcg, or 2000 mcg of folic acid once a day for 6 weeks
  Other Names: Folate
  Arms: 2; 3; 4; 5
Drug: Placebo Folic Acid — Placebo folic acid once a day for 6 weeks
  Arms: 1

SUMMARY:
High levels of homocysteine, which is an amino acid in the blood, have been linked to an increased risk of heart disease. This study will examine the effect that differing levels of folic acid have on reducing homocysteine levels among older adults.

DETAILED DESCRIPTION:
Elevated levels of homocysteine may be a risk factor for coronary heart disease, stroke, and peripheral vascular disease. Folate is a type of B vitamin that occurs naturally in food. In nutritional supplements, folate is known as folic acid, and it has been shown to lower the concentration of homocysteine in blood. Folic acid supplements are a simple way for people to increase their folate intake, lower their homocysteine levels, and reduce their risk of developing heart disease. However, more research is required to determine the most effective dose of folic acid needed to lower homocysteine levels. The purpose of this study is to examine the effect that varying doses of folic acid have on folate levels and homocysteine concentration levels in older adults.

This 6-week study will enroll healthy adults over the age of 60 who do not currently take multivitamins or B-vitamins. At a screening visit, participants will complete questionnaires on medical history, demographics, and diet. Also, height and weight will be measured, and a blood collection will occur. At a baseline study visit, participants will be randomly assigned to receive either placebo or one of four doses of folic acid-100 mcg, 400 mcg, 1000 mcg, or 2000 mcg-to be taken once a day for 6 weeks. Participants will attend a final study visit at Week 6, at which time another blood collection will occur.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Living in the Baltimore area

Exclusion Criteria:

* Taking multivitamins or B-vitamins
* Unwilling to discontinue supplements for 8 weeks before study entry
* Use of intramuscular vitamin B12
* Seizure disorder
* Pernicious anemia
* Long-term use of anti-folate drugs (e.g., methotrexate, sulfa-antibiotics)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 1996-06; Primary Completion 1996-09 (Actual); Study Completion 1996-09 (Actual)

PRIMARY OUTCOMES:
Plasma homocysteine levels | Measured at Week 6

SECONDARY OUTCOMES:
Serum folate levels | Measured at Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J. Appel, MD, MPH, Principal Investigator — Johns Hopkins University